CLINICAL TRIAL: NCT02015975
Title: Clinical Outcome After Treatment of Patellar Fractures With Locking Plates
Status: Completed | Type: Observational
Sponsor: Diakoniekrankenhaus Friederikenstift (Other)
Responsible Party: Sponsor
Other Study IDs: 001-2013
Record Dates: First submitted 2013-08-08; First posted 2013-12-19 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Fracture of Patella
Keywords: patellar fracture; fracture of patella; patella; locking plate osteosynthesis; osteosynthesis; star-plate; arrow-plate
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Depending on the fracture pattern of patellar fractures tension band wiring, interfragmentary screw fixation or combinations are common treatments. But there are several problems associated with these techniques as fracture dislocation or loosening and perforation of the wire. Furthermore an anatomic reduction with stable fixation in comminuted fractures is almost impossible to achieve.

A new option in the treatment of patellar fractures is the locking plate osteosynthesis, which provides a more stable fixation and higher mechanical strength in biomechanical tests compared to classic tension band wiring. Due to various screw positioning a stable fixation in comminuted fractures can be achieved and an early functional treatment with full weight bearing reduces the loss of knee-motion. Furthermore a removal of the osteosynthesis seems not to be essential anymore and the blood supply is not to be compromised.

Because of the absent of clinical evidence investigators want to evaluate the clinical outcome after locking plate osteosyntheses in patellar fractures and compare patient satisfaction, functional motion, complications and number of revisions with common treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients with indication for operative treatment of a patellar fracture
* sufficient compliance
* signed patient information

Exclusion Criteria:

* preoperative disease or trauma of the patellar
* preoperative loss of motion of the knee
* former operations of the patellar
* alcohol or drug consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a fracture of the patellar, which were operated with a locking plate osteosynthesis in the Friederikenstift Hannover since May 2013.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical short-term results | 6 weeks
  The clinical short-term results after treating a patellar fracture with plate osteosynthesis are evaluated. Therefore functional motion is measured, complications and revision operations reviewed and knee-scores analyzed (Tegner-Score, Lysholm-Score, Kujala-Score, International Knee Documentation Committee - Subjective knee evaluation form).

SECONDARY OUTCOMES:
Clinical long-term results | 24 months
  Further changes in functional motion and knee-scores are analyzed as well as the occurrence and frequency of complications and revision operations.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ellwein, Dr., Principal Investigator — Friederikenstift Hannover
Locations (1):
- Diakoniekrankenhaus Friederikenstift Hannover, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Ellwein A, Lill H, DeyHazra RO, Smith T, Katthagen JC. Outcomes after locked plating of displaced patella fractures: a prospective case series. Int Orthop. 2019 Dec;43(12):2807-2815. doi: 10.1007/s00264-019-04337-7. Epub 2019 Apr 30. PMID 31041522